CLINICAL TRIAL: NCT01672567
Title: Effects of Egg Ingestion on Endothelial Function in Adults With Coronary Artery Disease: A Randomized, Controlled, Crossover Trial
Brief Title: Effects of Egg Ingestion on Endothelial Function in Adults With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-05
Record Dates: First submitted 2011-08-09; First posted 2012-08-27 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Egg Consumption; Endothelial Function
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Egg supplementation (Experimental): Daily consumption of 2 eggs for breakfast for 6 weeks
  Interventions: Dietary Supplement: Egg supplementation
- Egg substitute (Experimental): Daily consumption of 1/2 cup of Egg Beater for breakfast for 6 weeks
  Interventions: Dietary Supplement: Egg substitute
- Control diet (Experimental): Daily consumption of high carbohydrate breakfast diet for 6 weeks, consisting of any of the following choices during each day of the treatment period: bagel, waffles, pancakes, or cereal and milk
  Interventions: Dietary Supplement: Control diet

INTERVENTIONS:
Dietary Supplement: Egg supplementation — Daily consumption of 2 eggs for breakfast for 6 weeks
  Arms: Egg supplementation
Dietary Supplement: Egg substitute — Daily consumption of 1/2 cup of Egg Beater for breakfast for 6 weeks
  Arms: Egg substitute
Dietary Supplement: Control diet — Daily consumption of high carbohydrate breakfast diet for 6 weeks, consisting of any of the following choices during each day of the treatment period: bagel, waffles, pancakes, or cereal and milk
  Arms: Control diet

SUMMARY:
The purpose of this study is to determine the effects of daily consumption of eggs or egg substitute for 6 weeks on endothelial function and on cholesterol and lipoprotein levels in participants with clinically established coronary heart disease (CHD).

DETAILED DESCRIPTION:
Restriction of dietary cholesterol, and thus the avoidance or restriction of egg intake, is routinely recommended to patients with coronary disease. However, the relative importance of dietary cholesterol to serum lipids has become a subject of active debate. Eggs provide a complete array of amino acids and an array of micronutrients, and are low in total fat. Epidemiological and clinical studies have showed that dietary intake of omega-3 fatty acids decreases the risk of coronary heart disease (CHD). Endothelial function testing represents a uniquely valuable means of assessing aggregated influences on cardiac risk by gauging physiologic responses of the vascular endothelium. In prior studies the investigators have shown that daily egg ingestion for 6 weeks did not adversely affect endothelial function in healthy adults or in hyperlipidemic adults. The investigators now propose a prospective, randomized, single-blind crossover study to assess the effects of eggs, egg substitute and high-carbohydrate American breakfast on endothelial responses and serum lipids in participants with clinically established CHD.

ELIGIBILITY:
Inclusion Criteria:

1. Males age greater than 35 years;
2. Post-menopausal females not currently on hormone replacement therapy;
3. Non-smokers;
4. CVD as defined by the presence of at least one coronary stenosis >50% determined angiographically or a documented history of myocardial infarction.

Exclusion Criteria:

1. Failure to meet inclusion criteria;
2. Anticipated inability to complete study protocol for any reason;
3. Current eating disorder;
4. Use of lipid-lowering or antihypertensive medications unless stable on medication for at least 3 months and willing to refrain from taking medication for 12 hours prior to EF scanning;
5. Regular use of high doses of vitamin E or C;
6. Use of insulin, glucose-sensitizing medication, vasoactive medication (including glucocorticoids, antineoplastic agents, psychoactive agents, or bronchodilators) or nutraceuticals;
7. Regular use of fiber supplements;
8. Diabetes;
9. Sleep apnea;
10. Restricted diets by choice (i.e., vegetarian, vegan);
11. Coagulopathy, known bleeding diathesis, or history of clinically significant hemorrhage; current use of warfarin.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Endothelial Function Flow mediated dilatation (FMD) as the percent change in brachial artery diameter from pre-cuff inflation to 60 seconds post-cuff release. | 6 weeks
  FMD will be measured as the percent change in brachial artery diameter from pre-cuff inflation to 60-seconds post-cuff release (upper arm cuff position). In addition to brachial diameter at 60 seconds post-cuff release, flow after cuff deflation within the first 15 seconds will be used as an indicator of stimulus strength, hyperemic flow being the stimulus for endothelial reactivity.

SECONDARY OUTCOMES:
Fasting Lipid Panel - Total cholesterol, low density lipoprotein cholesterol, high density lipoprotein cholesterol, triglyceride level, cholesterol / high density lipoprotein cholesterol ratio | 6 weeks
  Total cholesterol, low density lipoprotein cholesterol, high density lipoprotein cholesterol, triglyceride level, cholesterol / high density lipoprotein cholesterol ratio
3-Day Food Diary | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David L. Katz, MD, MPH, Principal Investigator — Yale-Griffin Prevention Research Center
Locations (1):
- Griffin Hospital, Derby, Connecticut, United States

REFERENCES:
- [Derived] Katz DL, Gnanaraj J, Treu JA, Ma Y, Kavak Y, Njike VY. Effects of egg ingestion on endothelial function in adults with coronary artery disease: a randomized, controlled, crossover trial. Am Heart J. 2015 Jan;169(1):162-9. doi: 10.1016/j.ahj.2014.10.001. Epub 2014 Oct 7. PMID 25497262